CLINICAL TRIAL: NCT05122962
Title: Pathophysiologic Mechanism for Arrhythmias and Impaired Aerobic Capacity in Tetralogy of Fallot and Other Congenital Heart Diseases
Acronym: PACT
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alexander C. Egbe, Principal Investigator, Mayo Clinic
Other Study IDs: 21-005062; R01HL158517 (NIH)
Record Dates: First submitted 2021-10-04; First posted 2021-11-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Tetralogy of Fallot; Congenital Heart Disease
MeSH Terms: conditions — Tetralogy of Fallot; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Remote Heart Rhythm Monitoring — We will be looking to see if remote heart rhythm monitoring for 30 days at baseline, 12, and 24 months, helps for early identification of adverse cardiac events.

SUMMARY:
This study is being done to determine the mechanism(s) contributing to the onset of symptoms (i.e. shortness of breath and/or palpitations) as well as changes in heart structure in patients with congenital heart disease (CHD)

ELIGIBILITY:
Inclusion Criteria:

* Moderate (or greater) PR based on quantitative Doppler echocardiography.
* Repaired TOF
* Congenital Heart Disease diagnosis including but not limited to Ebstein's anomaly, coarctation of the aorta (COA), Fontan palliation, transposition of the great arteries, congenitally corrected transposition of the great arteries.

Exclusion Criteria:

* Pregnant Women
* Unable to undergo CMRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a prospective study of patients with congenital heart disease receiving care at Mayo Clinic Rochester, MN.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Right Heart Remodeling | 24 Months
  Right Heart Remodeling measured via right atrial reservoir strain (%).

SECONDARY OUTCOMES:
Incident arrhythmias | 24 Months
  Incident of atrial flutter, atrial fibrillation, atrial tachycardia, and/or ventricular tachycardia.
Aerobic Capacity | 24 Months
  Aerobic Capacity measured as maximal oxygen consumption (ml/kg/min).

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Egbe, MBBS, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials